CLINICAL TRIAL: NCT01592630
Title: Effectiveness of Adding Transverse Abdominus Plane (TAP) Catheter Blocks to Patient-controlled Analgesia (PCA) in Laparoscopic Colon Resections: a Prospective, Randomized Controlled Study
Brief Title: Effectiveness of Transverse Abdominus Plane Catheter Blocks to Patient-controlled Analgesia in Laparoscopic Colon Resections
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Investigator Left Institution
Sponsor: Stamford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-1017.01
Record Dates: First submitted 2012-05-01; First posted 2012-05-07 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Colorectal Disorders; Observation of Neuromuscular Block
MeSH Terms: interventions — Ropivacaine; Drugs, Investigational; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Experimental): Subjects with TAP catheters attached to the On-Q pump with 0.2% ropivacaine
  Interventions: Drug: 0.2% ropivacaine
- Saline (Placebo Comparator): Subjects with TAP catheters attached to the On-Q pump with saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: 0.2% ropivacaine — On-Q pumps containing 0.2% ropivacaine to be attached to TAP catheters
  Other Names: Experimental drug
  Arms: Ropivacaine
Drug: Saline — On-Q pumps containing saline to be attached to TAP catheters
  Other Names: Control/Placebo
  Arms: Saline

SUMMARY:
The control of postoperative pain has become a major issue in surgery awareness and it is considered an important measurement of patient satisfaction. Improvements in pain relief, including stopping pain before it starts (i.e. preemptive treatment) is of great benefit to the surgical patient. When pain is aggressively addressed, patients respond by recovering faster.

The use of opioids remains the mainstay to minimize postoperative pain. Lately, long acting local anesthetic wound infiltration has been widely recognized as a useful adjunct to multimodal postoperative pain management. On that basis, a system that delivers a continuous local anesthetic to the surgical wound was developed, and better pain control has been achieved after several surgical procedures.

In patients undergoing abdominal procedures, such as colon resection, adequate pain control remains an issue. It is known that innervation to the antero-lateral abdomen is provided by sensory nerves T7-L1, ilioinguinal and iliohypogastric nerves, which travel through the transverse abdominis muscle plane (TAP). Local anesthetic block of these nerves has been described and has shown to be effective for immediate postoperative pain control.

Recently, the use of the On-Q pain relief system with catheters placed within the TAP has been evaluated. Published results have shown significant improvement of pain control (Forastiere). The idea of placing the pain catheters at the TAP plane seems to be more coherent with the anatomical distribution of the sensory nerves trunks. Due to the lack of prospective trials investigating the effectiveness of a continuous wound infusion with local anesthetics after general surgery procedures the investigators sought to determine the efficacy of this technique after laparoscopic colon resection procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 - 100 years of age undergoing laparoscopic colon resections.
* Patients must be able to read and write English.

Exclusion Criteria:

* Patients undergoing open procedures.
* Lap converted to open procedures.
* Patients with known liver dysfunction, or the following laboratory assays: ALT/AST/alk. Phos/total bilirubin of 2x ULN
* Cirrhosis Child's class A-C, INR >1.5. There is no specific isolated value of protein or albumin which would disqualify the subject.
* All emergent/urgent cases taken to the OR for colon resections.
* All patients with previous drug abuse/narcotic abuse history.
* Patients without the mental capacity to consent for the procedure/study.
* Subjects requiring a translator in order to sign the informed consent.
* Subjects with a history of an allergic reaction to local anesthetics or acetaminophen.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Time to flatus | 1 week
  Post-operative time measurement for the patient to pass flatus
Hospital Length of Stay | 1 week
  Post-operative time measurement until patient discharge

SECONDARY OUTCOMES:
Passage of Stool | 1 week
  Post-operative time measurement for the patient to pass stool
Narcotic use | 1 week
  Post-operative measurement of patient narcotic requirements

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Colon and Rectal Surgery, Stamford, Connecticut
  - Stamford Hospital, Stamford, Connecticut

REFERENCES:
- [Background] Gupta A, Fant F, Axelsson K, Sandblom D, Rykowski J, Johansson JE, Andersson SO. Postoperative analgesia after radical retropubic prostatectomy: a double-blind comparison between low thoracic epidural and patient-controlled intravenous analgesia. Anesthesiology. 2006 Oct;105(4):784-93. doi: 10.1097/00000542-200610000-00025. PMID 17006078
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Niraj G, Kelkar A, Jeyapalan I, Graff-Baker P, Williams O, Darbar A, Maheshwaran A, Powell R. Comparison of analgesic efficacy of subcostal transversus abdominis plane blocks with epidural analgesia following upper abdominal surgery. Anaesthesia. 2011 Jun;66(6):465-71. doi: 10.1111/j.1365-2044.2011.06700.x. Epub 2011 Apr 4. PMID 21457153
- [Background] Raue W, Haase O, Junghans T, Scharfenberg M, Muller JM, Schwenk W. 'Fast-track' multimodal rehabilitation program improves outcome after laparoscopic sigmoidectomy: a controlled prospective evaluation. Surg Endosc. 2004 Oct;18(10):1463-8. doi: 10.1007/s00464-003-9238-y. Epub 2004 Aug 26. PMID 15791370
- [Background] Chester JF, Ravindranath K, White BD, Shanahan D, Taylor RS, Lloyd-Williams K. Wound perfusion with bupivacaine: objective evidence for efficacy in postoperative pain relief. Ann R Coll Surg Engl. 1989 Nov;71(6):394-6. PMID 2604350
- [Background] Faucett J, Gordon N, Levine J. Differences in postoperative pain severity among four ethnic groups. J Pain Symptom Manage. 1994 Aug;9(6):383-9. doi: 10.1016/0885-3924(94)90175-9. PMID 7963791
- [Background] Edwards CL, Fillingim RB, Keefe F. Race, ethnicity and pain. Pain. 2001 Nov;94(2):133-137. doi: 10.1016/S0304-3959(01)00408-0. PMID 11690726
- [Background] De Oliveira GS Jr, Fitzgerald PC, Marcus RJ, Ahmad S, McCarthy RJ. A dose-ranging study of the effect of transversus abdominis block on postoperative quality of recovery and analgesia after outpatient laparoscopy. Anesth Analg. 2011 Nov;113(5):1218-25. doi: 10.1213/ANE.0b013e3182303a1a. Epub 2011 Sep 16. PMID 21926373